CLINICAL TRIAL: NCT01564108
Title: An Exploratory Study of Ranibizumab (Lucentis) for Treatment of Uveitic Patients With Refractory Cystoid Macular Oedema Which Has Proven Refractory or Ineligible to Standard Treatment.
Brief Title: The LIMO Study, Lucentis for Treatment of Uveitic Patients With Refractory Cystoid Macular Oedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OKHN1005
Record Dates: First submitted 2012-03-14; First posted 2012-03-27 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Uveitis Related Cystoid Macular Edema; Steroid-induced Glaucoma - Borderline
Keywords: Intravitreal Ranibizumab; Non-infectious uveitis; Refractory Cystoid Macular Oedema; Lucentis; LIMO
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental): Series of intravitreal injections of Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Series of intravitreal injections of Ranibizumab
  Other Names: Lucentis

SUMMARY:
Anti-vascular endothelial growth factor (VEGF) treatments show great promise in the treatment of a variety of retinal diseases. This study addresses a condition which affects a large number of our patients in whom the investigators face difficult management decisions. These patients with uveitis are severely disabled with visual loss related to cystoid macular oedema (CMO) and few options remain when standard treatment has either failed or is contraindicated.

The concentration of VEGF is increased in the eyes of patients with uveitis. Our hypothesis is that a series of injections of Ranibizumab may be an effective treatment for CMO. It is hoped that anti-VEGF therapy will have fewer side-effects than existing therapies and will be more effective in improving quality of life by reducing macular thickening and restoring visual function.

DETAILED DESCRIPTION:
The study has been designed as an open label, prospective non-randomised interventional case series.

Clinical staff will be asked to briefly discuss the option of enrolling into the study with potentially suitable patients. If the patient expresses an interest in finding out more about the study, the doctor will then contact a member of the study team, who will provide the patient with the patient information leaflet. This outlines the details and purpose of the study, the intended benefits of the intravitreal treatment and the potential hazards (including the unlicensed use of Ranibizumab for this indication). The intravitreal injection procedure will be discussed. The follow-up schedule will be outlined. There will be an opportunity for the patient to ask questions and at least 24 hours for the patient to think about entering the study. Only 1 eye of each patient, the worse eye, will be enrolled.

Comprehensive pre- and post- therapy and a longitudinal series of structure and function tests will be performed on all 20 enrolled patients. All patients will receive intravitreal injections performed in a designated clean room. The injections (Ranibizumab 0.5 mg in 0.05 ml) will be administered 4-5 weekly, for three injections then according to clinical need for a total of 12 months of follow-up. A maximum of 5 intravitreal Ranibizumab injections will be administered to patients who do not demonstrate any positive clinical response.

The patients will be seen for baseline screening over a 2 day period, with the first treatment with Ranibizumab administered on the second day (maximum of 10 working days after the first baseline screening day). Subsequent to the first 3 injections, the investigator will assess whether re-treatment is warranted (clinical / OCT criteria set out in re-treatment protocol). Re-treatment, when indicated, will be performed on the same day as the follow-up visit and no sooner than 4 weeks or later than 5 weeks from the time of the last treatment. If re-treatment with IVI Ranibizumab is to be deferred patients will not be given a sham injection. Should a relapse in ocular inflammation occur, it might be difficult to differentiate as to whether this is because of the drug or the underlying disease. A mild flare up, Lucentis-related or not, may be observed and treated with topical therapy (but patient will remain in the study). A moderate to severe recurrence, regardless of the cause which will necessitate more extensive therapy, namely a change or addition of systemic therapy, will result in the patient exiting the study-this would be an end point.

ELIGIBILITY:
Inclusion Criteria:

1. Cystoid macular oedema (CMO) from non-infectious uveitis:

   * Unilateral or Bilateral CMO (the worse eye only will be treated with intravitreal Ranibizumab) in a quiet eye for 1month.
   * On clinical exam and OCT, definite retinal thickening due to uveitic macular oedema involving the centre of the macula, refractory or ineligible for standard care.
   * Spectralis SD-OCT central subfield >=270 μm within 10 working days of study entry with uveitic macular oedema (cystoid or diffuse).
   * Quiet eye

     * as defined by 0-0.5 plus of cells in anterior chamber of the eye, and 0.5 or less vitreous haze (SUN classification).
     * topical / systemic immunosuppressive treatment allowed but stable for 2 month with no resolution of CMO in a quiet eye for 1 month.
     * greater than 3 months since orbital steroid injection, 4 months since intravitreal triamcinolone treatment, or 8 weeks since starting new oral therapy
     * at least 1 prior trial of oral, orbital or intravitreal steroid therapy for CMO or not eligible for steroid treatment (oral, orbital or intravitreal steroid) because IOP > 30 mmHg following such use in study eye or fellow eye (i.e. patient is a known steroid responder), at any time in the past.
2. Best corrected visual acuity in the study eye must be between 69 and 35 ETDRS letter score at 4m (Snellen equivalent of 6/12-6/60) within 10 working days of enrolment.

Exclusion Criteria:

1. Other causes of macular oedema e.g. diabetic macular oedema etc.
2. Presence of an ocular disease that in the opinion of the investigator is responsible for visual loss (e.g. sub-foveal atrophy, optic atrophy, dense subfoveal hard exudates).
3. Evidence of irreversible central visual loss
4. Evidence of visually significant vitreo-retinal traction or epiretinal membrane on OCT.
5. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e. cataract would be reducing acuity to 6/12 or worse if eye was otherwise normal).
6. History of cataract surgery within prior 6 months or cataract surgery anticipated within 6 months of starting the trial.
7. Any anti-VEGF treatment to study eye within 4 months.
8. Uncontrolled IOP > = 24 mmHg (on topical IOP lowering medications).
9. History of glaucoma.
10. Patients with active or suspected ocular or periocular infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The number of patients in whom, by consensus, no further treatment is required. | Data will be collected at every patient visit which will take place every 4-5 weeks, and analysed at 12 months follow-up
  Intravitreal Ranibizumab will be given at baseline, month 1 and month 2 . Subsequent 4-5 weekly injections will be given according to clinical need. There will be a total of 12 months of follow-up.
Change in CRT as measured by Spectralis spectral domain OCT. | at baseline visit then at 6 and 12 months.

SECONDARY OUTCOMES:
Functional vision changes based on self-reported quality of life measures (including acceptability of 4 weekly intravitreal therapy). | at baseline visit then at 6 and 12 months.
The proportion of subjects gaining >10 and >15 letters. | at baseline vist, on day 7 and day 14, then on monthly basis.
Change in contrast sensitivity. | at baseline visit then at months 1, 3, 6, 9 and 12.
Change in BCVA. | at baseline visit then at 3, 6, 9 and 12 months.
The proportion of subjects with loss of >15 letters and >30 letters. | at baseline vist, on day 7 and day 14, then on monthly basis.
Change in retinal sensitivity on microperimetry. | at baseline visit then on month 3, 6, 9 and 12.
Change in reading speed. | at baseline visit, months 1, 3,6, 9 and 12.
Evidence of improvement in PERG or mfERG. | at baseline visit, month 4, and 12.
Maintenance of the foveal avascular zone. | at baseline, 6 and 12.
Absence of toxicity on Electrophysiological testing / microperimetry / autofluorescence. | at baseline visit then on month 3, 4,6, 9 and 12.
Incidence and severity of ocular adverse events. | at day 7, day 14, month 1 then every month until 12 month post initial intravitreal injection
Incidence and severity of non ocular adverse events. | at day 7, day 14, month 1 then every month until 12 month post initial intravitreal injection

CONTACTS AND LOCATIONS:
Overall Officials: Narciss Okhravi, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHSFT Research and Treatment Centre, London, United Kingdom